CLINICAL TRIAL: NCT01149811
Title: A Randomized, Double-Blind, Crossover Study Comparing the Safety and Tolerability of Two Dose Regimens of Oromucosal Fipamezole ODT in Adult Patients With Parkinson's Disease Who Are Receiving Levodopa
Brief Title: A Study Comparing the Safety and Tolerability of Two Doses of Fipamezole in Adult Patients With Parkinson's Disease
Acronym: Fipamezole
Status: Completed | Type: Observational
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BVF-025-201
Record Dates: First submitted 2010-06-10; First posted 2010-06-24 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Parkinson's Disease
Keywords: Dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fipamezole ODT Cohort 1
  Interventions: Drug: Fipamezole ODT
- Fipamezole ODT Cohort 2
  Interventions: Drug: Fipamezole ODT Cohort 2

INTERVENTIONS:
Drug: Fipamezole ODT — Subjects will receive fipamezole ODT 15 mg three times daily for 1 week followed by fipamezole ODT 30 mg three times daily for 1 week, followed by a 2-week washout period. Beginning at Visit 5, subjects will receive fipamezole ODT 30 mg three times daily for 2 weeks.
  Groups: Fipamezole ODT Cohort 1
Drug: Fipamezole ODT Cohort 2 — Subjects will receive fipamezole ODT 30 mg three times daily for 2 weeks, followed by a 2-week washout period. Beginning at Visit 5, subjects will receive fipamezole ODT 15 mg three times daily for 1 week followed by fipamezole ODT 30 mg three times daily for 1 week.
  Groups: Fipamezole ODT Cohort 2

SUMMARY:
The purpose of this clinical trial is to compare the safety and tolerability of two dose regimens of fipamezole in adult patients with Parkinson's Disease who are receiving levodopa.

DETAILED DESCRIPTION:
Parkinson's Disease is the second most common neurodegenerative disorder worldwide. While treatment with dopaminergic agents like levodopa, the mainstay of treatment, is effective in the early phases of the disease, their benefits decrease with disease progression, and problems such as dyskinesia and on-off phenomenon begin to manifest. This study investigates the safety and tolerability of fipamezole at two dose levels in patients with Parkinson's Disease.

The sampling method used was simple random sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a man or woman between 30 and 75 years of age, inclusive, with intact oral mucosa at Screening (Visit 1) and Randomization (Visit 2).
2. Subject has a diagnosis of idiopathic Parkinson's disease defined according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnosis criteria.
3. Subject has been receiving a stable regimen of at least three daily administrations of levodopa (with a peripheral dopa decarboxylase inhibitor), with no dose changes for at least 4 weeks prior to Randomization (Visit 2).
4. Subject is rated at stage 2 to 4 on the Hoehn and Yahr scale.
5. If currently taking other medications (other than levodopa), subject must be on a stable regimen, defined as no dose changes for at least 1 month prior to Randomization (Visit 2).
6. Subject demonstrates the ability to comprehend the study procedures and provide informed consent.
7. Female subjects must be either postmenopausal for at least 1 year or surgically sterilized at least 3 months prior to Randomization (Visit 2). Male subjects must either be sterile or willing to use 2 approved methods of contraception when engaged in sexual intercourse with a female partner from Randomization (Visit 2) until 30 days after the last dose of study drug.

Exclusion Criteria:

1. Subject participated in an investigational medication study within the 3 months prior to Randomization (Visit 2).
2. Subject has immediate family members who are site Investigators or sponsor employees.
3. Subject has a history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or oncologic or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
4. Subject has impaired renal function (defined as a creatinine level of ≥ 1.5 times the upper limit of normal) at Screening (Visit 1).
5. Subject has impaired hepatic function (defined as SGOT/AST or SGPT/ALT levels ≥ 1.5 times the upper limit of normal) at Screening (Visit 1).
6. Subject has second- or third-degree atrioventricular block or sick sinus syndrome, atrial fibrillation, atrial flutter, severe or unstable angina, congestive heart failure, or myocardial infarction within 3 months of the screening visit or a significant ECG abnormality, including a QRS > 110 msec, a PR interval > 230 msec, a QTc ≥ 450 msec for male subjects, or a QTc ≥ 470 msec for female subjects.
7. Subject is at immediate risk of requiring hospitalization.
8. Subject has, in the opinion of the Investigator, a clinically important abnormality on his/her physical examination, electrocardiography, vital sign measurements, or laboratory assessment.
9. Subject is being treated with a disallowed medication that cannot be discontinued prior to Randomization (Visit 2) (see Table 5).
10. Subject has a current diagnosis of substance abuse or history of alcohol or drug abuse in the past 2 years prior to Screening (Visit 1).
11. Subject has positive findings on urine drug screen at Screening (Visit 1).
12. Subject has an allergy to fipamezole or the excipients.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease on stable regimen of levodopa
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To compare the safety and tolerability of two dose regimens of fipamezole orally disintegrating tablets (ODT) in adult patients with Parkinson's Disease who are receiving levodopa | Days -14 to 49
  Safety will be evaluated by assessing adverse events (AEs), vital signs (supine and orthostatic systolic and diastolic blood pressure, radial pulse rate), 12-lead ECG, blood and urine laboratory panels, and physical examination. Signs and symptoms of Parkinson's disease will be assessed using Hoehn and Yahr scale during the 'on' state.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph T. Doyle, Study Director — Bausch Health Americas, Inc.
Locations (4):
- United States (4):
  - CNS Network, Inc., Torrance, California
  - University of South Florida, Tampa, Florida
  - Advanced Neurodiagnostic Center, Metairie, Louisiana
  - Quest Research Institute, Bingham Farms, Michigan